CLINICAL TRIAL: NCT06740552
Title: Effect of Evolocumab on Non-culprit Coronary Lesions in Patients With Multivessel Disease Following Acute Myocardial Infarction: A Target Trial Emulation
Brief Title: Evolocumab in Patients With Multivessel Coronary Disease After Acute Myocardial Infarction: A Target Trial Emulation
Acronym: EVEREST
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Shenkang Hospital Development Center (Unknown); Tongji Hospital (Other); RenJi Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai General Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC2024CRI050
Record Dates: First submitted 2024-12-15; First posted 2024-12-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Multivessel Coronary Artery Disease; Acute Myocardial Infarction (AMI)
Keywords: evelocumab; non-culprit vessel; multivessel coronary artery disease; acute myocardial infarction; outcome; target trial emulation
MeSH Terms: interventions — evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- TTE cohort: The TTE cohort is the finally anlyzed population. The participates are enrolled upon meeting the inclusion/exclusion criteria.
  Interventions: Drug: Evolocumab; Drug: Lipid Lowering Medication

INTERVENTIONS:
Drug: Evolocumab — Evolocumab 140mg every two weeks
Drug: Lipid Lowering Medication — Any lipid lowering medication, including statin, ezetimibe, fibrates and etc.

SUMMARY:
The goal of this Target Trial Emulation (TTE) study is to evaluate the effect of evolocumab on clinical prognosis in patients with multivessel disease (MVD) following acute myocardial infarction (AMI) who have deferred non-culprit vessel. The main question it aims to answer is:

Does evolocumab lower risks of major adverse cardiovascular events (MACE) in patients with deferred non-culprit vessel after AMI?

DETAILED DESCRIPTION:
This study aims to investigate the potential prognostic benefits of evolocumab in patients with MVD after AMI at 2-year follow-up. The primary endpoint is MACE, defined as a composite of cardiac death, myocardial infarction, stroke, angina-driven coronary revascularization, and rehospitalization for heart failure. This is a multicentre, cohort-based TTE study and the target RCT is the FOURIER trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Acute myocardial infarction diagnosed at hospital admission;
* Multivessel coronary artery disease diagnosed at primary invasive coronary angiography;
* Culprit vessel successfully revascularized;
* At lease 1 non-culprit vessel with ≥50% stenosis and deferred at the opinion of the operator, and no staged revascularization within 6 months.

Exclusion Criteria:

* Cardiac shock, hemodynamically unstable, or severe heart failure (Killip IV)
* Any cardiac surgery within 6 weeks prior to screening;
* Moderate to severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m^2 at screening;
* Contraindication or allergy to iodinated contrast agent;
* Malignancy except non-melanoma skin cancers, cervical, or breast ductal carcinoma in situ within the last 5 years;
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed in short term.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a TTE study based on a multicentered, consecutive cohort of AMI patients from 2021 to 2022 at five 3rd-tier hospital in Shanghai. Patients who were diagnosed as AMI and refferred to primary invasive coronary angiography are consecutively enrolled in this cohort, regardless of revascularization treatment and lipid lowering strategy. The five hospitals are Zhongshan Hospital, Renji Hospital, Tongji Hospital, Shanghai General Hospital, and Shanghai Tenth People's Hospital.
Sampling Method: Probability Sample
Enrollment: 1862 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
MACE | 2 years
  A composite of cardiac death, myocardial infarction, and rehospitalization for heart failure.

SECONDARY OUTCOMES:
Death | 2 years
  All-cause death
Myocardial infarction | 2 years
  Myocardial infarction denotes the presence of acute myocardial injury detected by abnormal cardiac biomarkers in the setting of evidence of acute myocardial ischemia, according to the Fourth Universal Definition of Myocardial Infarction (2018).
Rehospitalization for heart failure | 2 years
  Readmissions due to symptoms from clinically diagnosed heart failure with or without reduced left ventricular ejection fraction.

OTHER OUTCOMES:
Landmark analysis at 30 days | 30 days
  MACE at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD is under protection and surveilliance of Shanghai Hospital Development Ceter.

REFERENCES:
- [Result] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224